CLINICAL TRIAL: NCT06642428
Title: Effect of Vitamin D Supplementation on the Efficacy and Adverse Effects of Neoadjuvant Therapy in Patients with Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Breast Disease Diagnosis and Treatment Center, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2024003
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Vitamin D; Neoadjuvant Therapy; Breast Cancer; Adverse Reaction; Efficacy; Chemotherapy
Keywords: Vitamin D; Breast Cancer; Adverse Reaction; Efficacy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant therapy + vitamin D2 (Experimental): Before the start of treatment and every 3 weeks thereafter, participants will receive injections of vitamin D2 at a dosage of 10 mg until the completion of neoadjuvant therapy. They will undergo the standard neoadjuvant regimen, which includes the 10 mg injection of vitamin D2 per cycle during the therapy. The dosage of neoadjuvant drugs may be tailored based on the physician's clinical judgment.
  Interventions: Drug: Neoadjuvant therapy + vitamin D2
- Neoadjuvant therapy (Other): Participants will receive the standard neoadjuvant regimen during each cycle of neoadjuvant therapy. The dosage of the neoadjuvant drugs may be tailored based on the physician's clinical judgment.
  Interventions: Drug: Neoadjuvant therapy

INTERVENTIONS:
Drug: Neoadjuvant therapy + vitamin D2 — Before the start of treatment and every 3 weeks thereafter, participants will receive injections of vitamin D2 at a dosage of 10 mg until the completion of neoadjuvant therapy. They will undergo the standard neoadjuvant regimen, which includes the 10 mg injection of vitamin D2 per cycle during the therapy. The dosage of neoadjuvant drugs may be tailored based on the physician's clinical judgment.
  Arms: Neoadjuvant therapy + vitamin D2
Drug: Neoadjuvant therapy — Participants will receive the standard neoadjuvant regimen during each cycle of neoadjuvant therapy. The dosage of the neoadjuvant drugs may be tailored based on the physician's clinical judgment.
  Arms: Neoadjuvant therapy

SUMMARY:
This randomized controlled Phase III trial was designed to evaluate the impact of supplemental vitamin D (VD) on the efficacy and side effects of neoadjuvant therapy in patients with breast cancer.

DETAILED DESCRIPTION:
This is a parallel-group, open-label randomized controlled trial designed to investigate the effects of supplemental vitamin D (VD) on the outcomes and side effects of neoadjuvant therapy in patients with breast cancer. Both groups will receive standard neoadjuvant therapy on day 1 and for each subsequent cycle. Additionally, vitamin D2 will be randomly administered to both groups.Blood samples and imaging results will be collected and analyzed prior to the initiation of neoadjuvant therapy and after every two cycles. Key outcomes to be recorded include the pathological complete response rate (pCR), objective response rate (ORR), disease control rate (DCR), and grade III or higher adverse effects related to neoadjuvant therapy. The primary and secondary study findings, along with adverse events, will be thoroughly evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
2. Primary diagnosis of breast cancer confirmed by preoperative pathological examination.
3. Serum 25(OH)D levels less than 20 ng/ml (50 nmol/L).
4. Patients who have not previously received chemotherapy and who plan to undergo at least 4 cycles of 5.neoadjuvant chemotherapy or combined targeted therapy.

6.Life expectancy of at least 6 months. 7.No other uncontrolled benign diseases at the time of recruitment. 8.All patients must have complete clinical medical records. 9.Willingness to voluntarily sign an informed consent form.

Exclusion Criteria:

1. History of invasive breast cancer.
2. Prior systemic treatment for the treatment or prevention of breast cancer.
3. Known allergic reactions to vitamin D or calcium compounds.
4. Comorbidities that may affect vitamin D or calcium balance or bone health.
5. Vitamin D or calcium supplementation in the past 3 months.
6. Presence of other tumors.
7. Pregnant or lactating women.
8. Individuals who do not wish to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The objective response rate | 4-6months
  Difference in change in the objective response rate from first to last assessment between two arms
The pathological complete response rate | 4-6months
  Difference in change the pathological complete response rate from first to last assessment between two arms

SECONDARY OUTCOMES:
The disease control rate | 4-6months
  Difference in change the disease control rate rate from first to last assessment between two arms
Evaluation of side effects related to neoadjuvant therapy (CTCAE v5.0). | From the initiation of neoadjuvant therapy to 21 days after the last cycle of neoadjuvant therapy.
  Side effects of neoadjuvant therapy will be assessed according to the CTCAE v5.0 criteria.
Pathological response assessment using the Miller & Payne scoring system in conjunction with residual disease in lymph nodes following neoadjuvant therapy. | 4-6months
  The pathological response will be assessed using the Miller & Payne scoring system, considering residual disease in lymph nodes after neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China